CLINICAL TRIAL: NCT00093964
Title: A Multicenter, Open-label, Randomized, Uncontrolled, Phase IIa Trial in Subjects With Recurrent Glioblastoma Multiforme to Investigate the Clinical Activity, Safety, and Tolerability of Cilengitide (EMD 121,974) Administered as a Single Agent.
Brief Title: Cilengitide (EMD 121974) for Recurrent Glioblastoma Multiforme (Brain Tumor)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMD 121974-009; NCT00103064 (obsolete NCT alias); NCT00119288 (obsolete NCT alias)
Record Dates: First submitted 2004-10-07; First posted 2004-10-11 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-01

CONDITIONS: Glioblastoma Multiforme
Keywords: Brain cancer; Brain tumor
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — Cilengitide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cilengitide 500 Milligram (mg) (Experimental)
  Interventions: Drug: Cilengitide 500 mg
- Cilengitide 2000 mg (Experimental)
  Interventions: Drug: Cilengitide 2000 mg

INTERVENTIONS:
Drug: Cilengitide 500 mg — Subjects will receive 1-hour intravenous infusion of 500 mg cilengitide twice weekly on Day 1 and 4 of each week during every 4-week cycle, for a total of 8 infusions per cycle. Cycles were repeated without pause until progressive disease (PD), unacceptable adverse events (AEs), or withdrawal of consent.
  Other Names: EMD 121974
  Arms: Cilengitide 500 Milligram (mg)
Drug: Cilengitide 2000 mg — Subjects will receive 1-hour intravenous infusion of 2000 mg cilengitide twice weekly on Day 1 and 4 of each week during every 4-week cycle, for a total of 8 infusions per cycle. Cycles were repeated without pause until progressive disease (PD), unacceptable adverse events (AEs), or withdrawal of consent.
  Other Names: EMD 121974
  Arms: Cilengitide 2000 mg

SUMMARY:
This study will investigate clinical activity, safety, and tolerability of the anti-angiogenic compound cilengitide (EMD 121974) in the treatment of first recurrence of glioblastoma multiforme (GBM).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained before undergoing any study-related activities.
* Males or females 18 years of age or older who can be treated in an outpatient setting.
* Histologically proven GBM, which is recurrent or progressive following surgery or biopsy, external beam radiation therapy, and 1 previous regimen of systemic chemotherapy (Gliadel wafer therapy is not considered systemic chemotherapy). Malignancy is to be documented with a previous histopathological report.
* Subjects initially diagnosed with other conditions similar to GBM (such as anaplastic astrocytoma [AA] or low grade glioma) that subsequently progressed to histologically proven GBM and have had surgery or biopsy, external beam radiation therapy, and 1 previous regimen of systemic chemotherapy for the original diagnosis are eligible if they meet all inclusion criteria.
* GBM recurring only in the contralateral hemisphere must be histologically confirmed by biopsy. GBM recurring bilaterally does not need to be histologically confirmed by biopsy (i.e., if recurrence is ipsilateral and contralateral).
* Archived tumor tissue specimens from the GBM surgery or biopsy must be available for central pathology review and exploratory analysis of angiogenic markers (e.g. αvβ3 and αvβ5 integrins).
* Measurable disease (solid contrast-enhancing lesion greater than or equal to (>=)1 cm in any dimension) evaluated by gadolinium-enhanced magnetic resonance imaging (Gd MRI) within 2 weeks prior to the first dose of EMD 121974.
* At least 12 weeks have elapsed since the last radiation treatment, and at least 4 weeks have elapsed since the last chemotherapy dose (at least 6 weeks for nitrosourea-containing chemotherapy) prior to the first dose of EMD 121974.
* If the subject underwent recent surgery, status must be >=2 weeks post surgery or >=1 week post biopsy, in stable condition, and maintained on a stable corticosteroid regimen for >=5 days prior to first dose of EMD 121974.
* Karnofsky Performance Score (KPS) of >=70%.
* Subjects with the potential for pregnancy or impregnating their partner must agree to follow acceptable methods of birth control to avoid conception during the study and for at least 6 months after receiving the last dose of study drug.
* Women of childbearing potential must have a negative pregnancy test at screening.
* Laboratory values (within 1 week prior to the first dose of EMD 121974, except for blood count and Prothrombin time (PT)/Partial thromboplastin time (PTT), which are to be within 72 hours of the first dose): Absolute neutrophil count >=1500/millimeter (mm)^3. Platelets >=100,000/mm^3. Creatinine less than or equal to (<=) 1.5 milligram/deciliter (mg/dL) or creatinine clearance >=60 mL/min. Hematocrit >=30%. Prothrombin time (PT) and partial thromboplastin time (PTT) within normal limits. Hemoglobin >=10 mg/dL. Total bilirubin <=1.5 times the upper limit of normal. Aspartate aminotransferase and alanine aminotransferase <=2.5 times above upper limit of normal.
* No more than 8 weeks have elapsed since recurrence was detected

Exclusion Criteria:

* Prior radiation therapy greater than (>) 66 Gray.
* Subject anticipates undergoing elective surgery, dental extraction, or invasive dental procedures.
* History of recent peptic ulcer disease (endoscopically proven gastric ulcer, duodenal ulcer, or esophageal ulcer) within 6 months of enrollment.
* History of prior malignancy. Subjects with curatively treated cervical carcinoma in situ or basal cell carcinoma of the skin, or subjects who have been free of other malignancies for ≥5 years are eligible for this study.
* History of coagulation disorder associated with bleeding or recurrent thrombotic events.
* Concurrent illness, including severe infection, which may jeopardize the ability of the subject to receive the procedures outlined in this protocol with reasonable safety.
* Subject is pregnant, anticipates becoming pregnant within 6 months after study participation, or is currently breast-feeding.
* Receiving concurrent investigational agents or has received an investigational agent within the past 30 days prior to the first dose of EMD 121974.
* Prior antiangiogenic therapy.
* Placement of Gliadel wafer at surgery for recurrence.
* Unable to undergo Gd MRI.
* Current known alcohol dependence or drug abuse.
* Requiring concomitant chemotherapy.
* Treatment with a prohibited concomitant medication.
* Known hypersensitivity to the study treatment.
* Legal incapacity or limited legal capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2004-10-13 (Actual); Primary Completion 2005-10-28 (Actual); Study Completion 2010-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Inc., a business of Merck KGaA, Darmstadt, Germany
Locations (17):
- United States (17):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Barrow Neurological Institute, Phoenix, Arizona
  - UCLA Medical Center, Los Angeles, California
  - Denise Damek, Aurora, Colorado
  - Northwestern University, Chicago, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Good Samaritan Hospital/Tri Health Hatton Center, Cincinnati, Ohio
  - Baylor University Medical Center at Dallas, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Vermont/Fletcher Allen Healthcare, Burlington, Vermont
  - University of Virginia Health System, Charlottesville, Virginia

REFERENCES:
- [Result] Reardon DA, Fink KL, Mikkelsen T, Cloughesy TF, O'Neill A, Plotkin S, Glantz M, Ravin P, Raizer JJ, Rich KM, Schiff D, Shapiro WR, Burdette-Radoux S, Dropcho EJ, Wittemer SM, Nippgen J, Picard M, Nabors LB. Randomized phase II study of cilengitide, an integrin-targeting arginine-glycine-aspartic acid peptide, in recurrent glioblastoma multiforme. J Clin Oncol. 2008 Dec 1;26(34):5610-7. doi: 10.1200/JCO.2008.16.7510. Epub 2008 Nov 3. PMID 18981465

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/Last subject in: 13 October 2004/28 October 2005. Data analysis cut-off: 21 October 2010
Groups:
- Cilengitide 500 Milligram (mg): Subjects received 1-hour intravenous infusion of 500 mg cilengitide twice weekly on Day 1 and 4 of each week during every 4-week cycle, for a total of 8 infusions per cycle. Cycles were repeated without pause until progressive disease (PD), unacceptable adverse events (AEs), or withdrawal of consent.
- Cilengitide 2000 mg: Subjects received 1-hour intravenous infusion of 2000 mg cilengitide twice weekly on Day 1 and 4 of each week during every 4-week cycle, for a total of 8 infusions per cycle. Cycles were repeated without pause until progressive disease (PD), unacceptable adverse events (AEs), or withdrawal of consent.
Period: Overall Study
Arm/Group | Cilengitide 500 Milligram (mg) | Cilengitide 2000 mg
Started | 41 | 40
Completed | 41 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cilengitide 500 Milligrams (mg): Subjects received a 1-hour intravenous (i.v.) infusion of 500 mg cilengitide twice weekly on Days 1 and 4 of each week during every 4-week cycle, for a total of 8 infusions per cycle. Cycles were repeated without pause until progressive disease (PD), unacceptable adverse events (AEs), or withdrawal of consent.
- Cilengitide 2000 mg: Subjects received a 1-hour intravenous (i.v.) infusion of 2000 mg cilengitide twice weekly on Days 1 and 4 of each week during every 4-week cycle, for a total of 8 infusions per cycle. Cycles were repeated without pause until progressive disease (PD), unacceptable adverse events (AEs), or withdrawal of consent.
- Total: Total of all reporting groups
Arm/Group | Cilengitide 500 Milligrams (mg) | Cilengitide 2000 mg | Total
Number analyzed (Participants) | 41 | 40 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (12.11) | 54.6 (11.4) | 53.8 (11.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 12 | 30
  Male | 23 | 28 | 51

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Progression-free Survival
Description: Progression-free survival was defined as subjects who survived greater than or equal to (>=) 180 days without disease progression. Disease progression was assessed as per independent central blinded radiology assessment.
Time Frame: Month 6
Population: The intention-to-treat (ITT) population included all randomized subjects who had received at least 1 intravenous administration of cilengitide. Here,"Number of participants analyzed" signifies those subjects who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Cilengitide 500 Milligrams (mg) | Cilengitide 2000 mg
Number analyzed (Participants) | 40 | 40
percentage of subjects | 7.5 [1.6 to 20.4] | 15.0 [5.7 to 29.8]

2. Secondary Outcome: Percentage of Subjects With Overall Response Rate
Description: Overall response rate was defined as percentage of subjects who had best response during the study which was either complete response (CR: disappearance of all tumors, no new lesions and stable or improved neurological examination) or partial response (PR: >= reduction in the sum of the products of the largest perpendicular diameters compared to the baseline sum, no worsening of evaluable lesion and stable or improved neurological examination). CR or PR was confirmed within 31 days with a repeat neuroimaging.
Time Frame: From the start of treatment up to 6 years
Population: ITT population included all randomized subjects who had received at least 1 intravenous administration of cilengitide. Here,"Number of participants analysed" signifies those subjects who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Cilengitide 500 Milligrams (mg) | Cilengitide 2000 mg
Number analyzed (Participants) | 40 | 40
percentage of subjects | 5.0 [0.6 to 16.9] | 12.5 [4.2 to 26.8]

3. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression was defined as the number of days between the first dose and the date of first assessment of progressive disease during the study or until death. Surviving subjects without progressive disease were censored at the time of the last visit and the subject was known to be non-progressing. Disease progression was assessed as per independent central blinded radiology assessment.
Time Frame: From the start of treatment until disease progression (assessed up to a maximum of 6 years)
Population: ITT population included all randomized subjects who had received at least 1 intravenous administration of cilengitide.
Measure: Median (Full Range); unit: months
Arm/Group | Cilengitide 500 Milligrams (mg) | Cilengitide 2000 mg
Number analyzed (Participants) | 41 | 40
months | 1.81 [0.39 to 56.71] | 1.91 [0.66 to 57.76]

4. Secondary Outcome: Overall Survival Time
Description: Survival time was defined as the number of months between the date of randomization and the date of death or the last date the subject was known to be alive.
Time Frame: From the start of treatment until death (assessed up to a maximum of 6 years)
Population: ITT population included all randomized subjects who had received at least 1 intravenous administration of cilengitide.
Measure: Median (Full Range); unit: months
Arm/Group | Cilengitide 500 Milligrams (mg) | Cilengitide 2000 mg
Number analyzed (Participants) | 41 | 40
months | 6.54 [1.45 to 65.92] | 9.91 [0.92 to 67.23]

5. Secondary Outcome: Percentage of Subjects With 1-year of Survival Rate
Description: 1-year survival rate was defined as percentage of subjects who survived for >=365 days with or without disease progression. Disease progression was assessed as per independent central blinded radiology assessment.
Time Frame: From the start of treatment up to 1 year
Population: ITT population included all randomized subjects who had received at least 1 intravenous administration of cilengitide.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Cilengitide 500 Milligrams (mg) | Cilengitide 2000 mg
Number analyzed (Participants) | 41 | 40
percentage of subjects | 22.0 [10.9 to 35.5] | 37.5 [22.9 to 52.1]

6. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Cmax is the maximum observed plasma concentration of cilengitide after administration.
Time Frame: Pre-dose, 1, 1.5, 2, 3, 4, 8, 24 hours post-infusion on Day 1 of Week 1 in Cycle 1 and 2
Population: The pharmacokinetic (PK) population: subjects who had received cilengitide and who had blood samples drawn in Week 1 that provided drug concentration for non-compartmental PK evaluation. Here,"Overall Number of participants analyzed" = subjects evaluable for this outcome and "Number analyzed" = subjects evaluable for the specified category.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | Cilengitide 500 Milligrams (mg) | Cilengitide 2000 mg
Number analyzed (Participants) | 5 | 6
microgram per milliliter (mcg/mL)
  Cycle 1: number analyzed (Participants) | 2 | 3
  Cycle 1 | 40.4 (24.4) | 105.7 (14.1)
  Cycle 2: number analyzed (Participants) | 3 | 3
  Cycle 2 | 35.4 (20.6) | 169.7 (20.7)

7. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax)
Description: Tmax is the time to reach the maximum plasma concentration (Cmax) of cilengitide.
Time Frame: Pre-dose,1,1.5,2,3,4,8 and 24 hours post-infusion on Day 1 of Week 1 in Cycles 1 and 2
Population: The PK population: subjects who had received cilengitide and who had blood samples drawn in Week 1 that provided drug concentration for non-compartmental PK evaluation. Here,"Overall Number of participants analyzed" = subjects evaluable for this outcome and "Number analyzed" = subjects evaluable for the specified category.
Measure: Median (Full Range); unit: Hour (h)
Arm/Group | Cilengitide 500 Milligrams (mg) | Cilengitide 2000 mg
Number analyzed (Participants) | 5 | 6
Hour (h)
  Cycle 1: number analyzed (Participants) | 2 | 3
  Cycle 1 | 1.13 [1.08 to 1.17] | 1.33 [1.08 to 1.50]
  Cycle 2: number analyzed (Participants) | 3 | 3
  Cycle 2 | 1.17 [1.08 to 1.25] | 1.00 [1.00 to 1.08]

8. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity After Administration (AUC 0-infinity)
Description: AUC 0-infinity is the area under the curve for the plot showing plasma concentration against time from time zero to the time of the last quantifiable concentration of cilengitide.
Time Frame: Pre-dose,1,1.5,2,3,4,8 and 24 hours post-infusion on Day 1 of Week 1 in Cycles 1 and 2
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Microgram per milliliter*hour (mcg/mL*h)
Arm/Group | Cilengitide 500 Milligrams (mg) | Cilengitide 2000 mg
Number analyzed (Participants) | 5 | 6
Microgram per milliliter*hour (mcg/mL*h)
  Cycle 1: number analyzed (Participants) | 2 | 3
  Cycle 1 | 92.7 (60.4) | 346.5 (50.3)
  Cycle 2: number analyzed (Participants) | 3 | 3
  Cycle 2 | 84.6 (33.2) | 429.3 (27.4)

9. Secondary Outcome: Apparent Terminal Rate Constant (Lambda z)
Description: Lambda z was determined from the terminal slope of the log-transformed plasma concentration curve using linear regression on terminal data points of the curve.
Time Frame: Pre-dose,1,1.5,2,3,4,8 and 24 hours post-infusion on Day 1 of Week 1 in Cycles 1 and 2
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Per hour (/h)
Arm/Group | Cilengitide 500 Milligrams (mg) | Cilengitide 2000 mg
Number analyzed (Participants) | 5 | 6
Per hour (/h)
  Cycle 1: number analyzed (Participants) | 2 | 3
  Cycle 1 | 0.320 (0.080) | 0.204 (0.010)
  Cycle 2: number analyzed (Participants) | 3 | 3
  Cycle 2 | 0.325 (0.107) | 0.211 (0.008)

10. Secondary Outcome: Terminal Half-life (t1/2)
Description: The t1/2 is the time taken to eliminate half the amount of cilengitide.
Time Frame: Pre-dose,1,1.5,2,3,4,8 and 24 hours post-infusion on Day 1 of Week 1 in Cycles 1 and 2
Population: as for outcome 7
Measure: Median (Full Range); unit: Hour (h)
Arm/Group | Cilengitide 500 Milligrams (mg) | Cilengitide 2000 mg
Number analyzed (Participants) | 5 | 6
Hour (h)
  Cycle 1: number analyzed (Participants) | 2 | 3
  Cycle 1 | 2.24 [1.84 to 2.63] | 3.38 [3.24 to 3.59]
  Cycle 2: number analyzed (Participants) | 3 | 3
  Cycle 2 | 2.04 [1.63 to 3.28] | 3.21 [3.21 to 3.42]

11. Secondary Outcome: Mean Residence Time of Drug in the Body (MRT)
Description: MRT is defined as the mean duration of time a drug molecule is present in the systemic circulation.
Time Frame: Pre-dose,1,1.5,2,3,4,8 and 24 hours post-infusion on Day 1 of Week 1 in Cycles 1 and 2
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Hour (h)
Arm/Group | Cilengitide 500 Milligrams (mg) | Cilengitide 2000 mg
Number analyzed (Participants) | 5 | 6
Hour (h)
  Cycle 1: number analyzed (Participants) | 2 | 3
  Cycle 1 | 2.76 (0.66) | 3.98 (0.25)
  Cycle 2: number analyzed (Participants) | 3 | 3
  Cycle 2 | 2.92 (0.74) | 3.42 (0.18)

12. Secondary Outcome: Total Body Clearance (CL) of Drug From Plasma/Cerebro Spinal Fluid (CSF)
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body, calculated as dose divided by AUC0-infinity.
Time Frame: Pre-dose,1,1.5,2,3,4,8 and 24 hours post-infusion on Day 1 of Week 1 in Cycles 1 and 2
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Liter per hour (L/h)
Arm/Group | Cilengitide 500 Milligrams (mg) | Cilengitide 2000 mg
Number analyzed (Participants) | 5 | 6
Liter per hour (L/h)
  Cycle 1: number analyzed (Participants) | 2 | 3
  Cycle 1 | 6.85 (4.47) | 5.85 (0.86)
  Cycle 2: number analyzed (Participants) | 3 | 3
  Cycle 2 | 6.75 (3.25) | 4.67 (0.31)

13. Secondary Outcome: Apparent Volume of Distribution During the Terminal Phase (Vz)
Description: Vz was calculated as Dose/(AUC0-infinity multiplied by elimination rate constant [lambda z]) following single dose.
Time Frame: Pre-dose,1,1.5,2,3,4,8 and 24 hours post-infusion on Day 1 of Week 1 in Cycles 1 and 2
Population: The PK population included the subjects who had received cilengitide and who had had blood samples drawn in Week 1 and/or 5 that provided drug concentration for non-compartmental PK evaluation. Here, "Number of participants analysed" signifies those subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Liter (L)
Arm/Group | Cilengitide 500 Milligrams (mg) | Cilengitide 2000 mg
Number analyzed (Participants) | 5 | 6
Liter (L)
  Cycle 1: number analyzed (Participants) | 2 | 3
  Cycle 1 | 20.3 (8.9) | 28.9 (5.5)
  Cycle 2: number analyzed (Participants) | 3 | 3
  Cycle 2 | 21.0 (6.8) | 22.1 (1.2)

14. Secondary Outcome: Apparent Volume of Distribution at Steady State (Vss)
Description: Vss is the theoretical volume that the total amount of administered drug would have to occupy (if it were uniformly distributed), to provide the same concentration as it is in blood plasma at steady state.
Time Frame: Pre-dose, 1, 1.5, 2, 3, 4, 8, 24 hours post-infusion on Day 1 of Week 1 in Cycle 1 and 2
Population: The PK population included the subjects who had received cilengitide and who had blood samples drawn in Week 1 and/or 5 that provided drug concentration for non-compartmental PK evaluation. Here, "Number of participants analysed" signifies those subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Liter (L)
Arm/Group | Cilengitide 500 Milligrams (mg) | Cilengitide 2000 mg
Number analyzed (Participants) | 5 | 6
Liter (L)
  Cycle 1: number analyzed (Participants) | 2 | 3
  Cycle 1 | 17.4 (7.8) | 23.3 (4.1)
  Cycle 2: number analyzed (Participants) | 3 | 3
  Cycle 2 | 19.3 (8.3) | 15.9 (0.9)

15. Secondary Outcome: Number of Subjects With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a subject which did not necessarily have a causal relationship with the study drug. A TEAE was any AE that started on or any time after the day of first dose of cilengitide during the treatment phase or within the safety follow-up after last dose of cilengitide. A SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening; persistent or significant disability/incapacity; congenital anomaly.
Time Frame: From the start of treatment up to 6 years
Population: The safety population included all randomized subjects who had received at least 1 intravenous administration of cilengitide.
Measure: Number; unit: subjects
Arm/Group | Cilengitide 500 Milligram (mg) | Cilengitide 2000 mg
Number analyzed (Participants) | 41 | 40
subjects
  TEAEs | 41 | 39
  SAEs | 16 | 18

ADVERSE EVENTS:
Arm/Group | Cilengitide 500 Milligram (mg) | Cilengitide 2000 mg
Serious Adverse Events (participants affected / at risk) | 16/41 | 18/40
Other Adverse Events (participants affected / at risk) | 41/41 | 39/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cilengitide 500 Milligram (mg) (N=41) | Cilengitide 2000 mg (N=40)
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Splenic artery aneurysm (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 2 | 1
Chest pain (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 1
Gait disturbance (General disorders) | 0 | 1
Generalised oedema (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Aspergillosis (Infections and infestations) | 0 | 1
Brain abscess (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1
Clostridium colitis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 0
Blood glucose increased (Investigations) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0
Aphasia (Nervous system disorders) | 2 | 3
Ataxia (Nervous system disorders) | 1 | 1
Brain oedema (Nervous system disorders) | 2 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 5 | 8
Grand mal convulsion (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 5 | 2
Hemiparesis (Nervous system disorders) | 1 | 1
Hemiplegia (Nervous system disorders) | 1 | 0
Motor dysfunction (Nervous system disorders) | 1 | 0
Neurologic neglect syndrome (Nervous system disorders) | 0 | 1
Neuropathy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Postictal paralysis (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Affective disorder (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 2 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cilengitide 500 Milligram (mg) (N=41) | Cilengitide 2000 mg (N=40)
Haemoglobinaemia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 2 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Deafness (Ear and labyrinth disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 2 | 2
Middle ear effusion (Ear and labyrinth disorders) | 1 | 0
Otorrhoea (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 1
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Cushingoid (Endocrine disorders) | 5 | 3
Hirsutism (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 1 | 1
Diplopia (Eye disorders) | 1 | 2
Dry eye (Eye disorders) | 1 | 0
Eye irritation (Eye disorders) | 1 | 0
Eye pain (Eye disorders) | 0 | 1
Eyelid oedema (Eye disorders) | 0 | 1
Gaze palsy (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 0 | 1
Lacrimation increased (Eye disorders) | 1 | 0
Ophthalmoplegia (Eye disorders) | 1 | 0
Papilloedema (Eye disorders) | 1 | 1
Photophobia (Eye disorders) | 1 | 0
Scleral haemorrhage (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 5 | 3
Visual acuity reduced (Eye disorders) | 5 | 1
Vitreous floaters (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Chapped lips (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 7 | 5
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 1
Faecal incontinence (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 3 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Gingival hypertrophy (Gastrointestinal disorders) | 1 | 0
Gingivitis (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 1
Lip disorder (Gastrointestinal disorders) | 0 | 1
Lip dry (Gastrointestinal disorders) | 0 | 1
Loose stools (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 10 | 6
Stomach discomfort (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 2
Abasia (General disorders) | 1 | 0
Adverse drug reaction (General disorders) | 1 | 0
Asthenia (General disorders) | 1 | 6
Catheter related complication (General disorders) | 0 | 1
Catheter site haemorrhage (General disorders) | 2 | 0
Catheter site oedema (General disorders) | 1 | 0
Catheter site pain (General disorders) | 1 | 2
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Chills (General disorders) | 1 | 1
Cyst (General disorders) | 0 | 2
Difficulty in walking (General disorders) | 1 | 1
Facial pain (General disorders) | 0 | 1
Fatigue (General disorders) | 11 | 18
Gait disturbance (General disorders) | 4 | 6
Influenza like illness (General disorders) | 1 | 0
Infusion site pain (General disorders) | 0 | 1
Infusion site reaction (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 12 | 10
Pitting oedema (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 3
Temperature intolerance (General disorders) | 1 | 1
Venipuncture site bruise (General disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 1
Seasonal allergy (Immune system disorders) | 2 | 0
Bacteriuria (Infections and infestations) | 1 | 0
Body tinea (Infections and infestations) | 1 | 0
Candidiasis (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 1 | 2
Conjunctivitis infective (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Dental caries (Infections and infestations) | 1 | 0
Eczema infected (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Eye infection (Infections and infestations) | 1 | 1
Folliculitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 0
Herpes simplex (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Hordeolum (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 1
Oral infection (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Sialoadenitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 3 | 2
Tooth abscess (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 2
Urinary tract infection (Infections and infestations) | 4 | 3
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 1
Blood blister (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 3 | 3
Excoriation (Injury, poisoning and procedural complications) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 6 | 3
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1
Post procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 3
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Tooth injury (Injury, poisoning and procedural complications) | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Activated partial thromboplastin time shortened (Investigations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 2
Anticonvulsant drug level increased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 2
Bacteria urine (Investigations) | 3 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 1
Blood cholesterol increased (Investigations) | 2 | 1
Blood glucose increased (Investigations) | 1 | 0
Blood iron decreased (Investigations) | 1 | 0
Blood potassium decreased (Investigations) | 0 | 1
Blood urea increased (Investigations) | 2 | 0
Cardiac murmur (Investigations) | 0 | 1
Electrocardiogram ST segment elevation (Investigations) | 1 | 0
Electrocardiogram abnormal (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1
Neutrophil count increased (Investigations) | 2 | 0
Nuclear magnetic resonance imaging abnormal (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Prothrombin time (Investigations) | 0 | 1
Red blood cell count decreased (Investigations) | 1 | 0
Tandem gait test abnormal (Investigations) | 1 | 1
Weight decreased (Investigations) | 0 | 1
Weight increased (Investigations) | 1 | 2
White blood cell count decreased (Investigations) | 0 | 1
White blood cells urine positive (Investigations) | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1
Markedly reduced dietary intake (Metabolism and nutrition disorders) | 1 | 0
Tetany (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle cramp (Musculoskeletal and connective tissue disorders) | 2 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Myopathy steroid (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 2
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Amnesia (Nervous system disorders) | 8 | 5
Aphasia (Nervous system disorders) | 5 | 9
Ataxia (Nervous system disorders) | 1 | 3
Aura (Nervous system disorders) | 2 | 0
Balance disorder (Nervous system disorders) | 7 | 2
Brain oedema (Nervous system disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 2 | 1
Convulsion (Nervous system disorders) | 7 | 4
Coordination abnormal (Nervous system disorders) | 2 | 1
Cranial nerve disorder (Nervous system disorders) | 1 | 2
Cranial neuropathy (Nervous system disorders) | 3 | 1
Disturbance in attention (Nervous system disorders) | 3 | 0
Dizziness (Nervous system disorders) | 7 | 7
Dysarthria (Nervous system disorders) | 3 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Dysgraphia (Nervous system disorders) | 0 | 1
Dyskinesia (Nervous system disorders) | 0 | 1
Dysphasia (Nervous system disorders) | 0 | 1
Facial palsy (Nervous system disorders) | 1 | 3
Facial paresis (Nervous system disorders) | 5 | 0
Grand mal convulsion (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 14 | 14
Hemianopia homonymous (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 3 | 4
Hemiplegia (Nervous system disorders) | 1 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 1
Hyperreflexia (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 2 | 2
Lethargy (Nervous system disorders) | 2 | 1
Memory impairment (Nervous system disorders) | 4 | 5
Motor dysfunction (Nervous system disorders) | 4 | 2
Neurologic neglect syndrome (Nervous system disorders) | 2 | 1
Neuropathic pain (Nervous system disorders) | 0 | 1
Neuropathy (Nervous system disorders) | 2 | 0
Nystagmus (Nervous system disorders) | 1 | 2
Paraesthesia (Nervous system disorders) | 2 | 2
Partial seizures (Nervous system disorders) | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 3
Peroneal nerve palsy (Nervous system disorders) | 0 | 1
Pyramidal tract syndrome (Nervous system disorders) | 1 | 0
Reflex sympathetic dystrophy (Nervous system disorders) | 1 | 0
Sensory disturbance (Nervous system disorders) | 1 | 1
Simple partial seizures (Nervous system disorders) | 1 | 2
Sinus headache (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 2
Speech disorder (Nervous system disorders) | 4 | 3
Tremor (Nervous system disorders) | 4 | 4
Upper motor neurone lesion (Nervous system disorders) | 2 | 0
Visual field defect (Nervous system disorders) | 1 | 0
Affect lability (Psychiatric disorders) | 1 | 1
Aggression (Psychiatric disorders) | 0 | 1
Agitation (Psychiatric disorders) | 2 | 1
Anxiety (Psychiatric disorders) | 2 | 3
Cognitive deterioration (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 8 | 7
Depression (Psychiatric disorders) | 3 | 6
Disorientation (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 4 | 6
Irritability (Psychiatric disorders) | 2 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Mood altered (Psychiatric disorders) | 2 | 1
Nervousness (Psychiatric disorders) | 1 | 0
Personality change (Psychiatric disorders) | 1 | 2
Psychomotor retardation (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 1
Leukocyturia (Renal and urinary disorders) | 1 | 0
Micturition urgency (Renal and urinary disorders) | 2 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 1
Pollakiuria (Renal and urinary disorders) | 2 | 0
Proteinuria (Renal and urinary disorders) | 4 | 0
Renal salt-wasting syndrome (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 4 | 4
Breast pain (Reproductive system and breast disorders) | 1 | 0
Menstrual disorder (Reproductive system and breast disorders) | 1 | 0
Nipple pain (Reproductive system and breast disorders) | 0 | 1
Polymenorrhoea (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Sexual dysfunction (Reproductive system and breast disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Face oedema (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 6 | 7
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1
Skin fragility (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 2
Petechiae (Vascular disorders) | 2 | 1
Phlebitis (Vascular disorders) | 0 | 1
Phlebitis superficial (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other